CLINICAL TRIAL: NCT02422342
Title: Comparison Study of Non-invasive Measurement of Blood Pressure and Cardiac Output During Stress Echocardiography
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HeartBeat Technologies LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: HeartBeat_V2.0_SE
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: High Cardiac Output; Low Cardiac Output
MeSH Terms: conditions — Cardiac Output, High; Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulse Oximeter CMS50FW (Contec Medical) — The patients will be wearing the pulse oximeter during the test period (20-30 minutes).
  The data from the oximeter will be sent by Bluetooth to the mobile application

SUMMARY:
The objectives of the clinical trial is to validate hemodynamic parameters (Blood pressure and Cardiac Output) generated by an application coupled with an off-the-shelf pulse oximeter. The validation will be done by comparing the generated information to data gathered while performing Stress Echocardiography. The first phase of the study will be done on 10 patients undergoing a Stress Echocardiography test at the cardiology department at Meir Hospital

DETAILED DESCRIPTION:
The HeartBeat system combines an FDA/CE approved watch-like Pulse Oximeter for acquiring the data and an android software application that serves as the Hemodynamic calculator. The application performs POST-PROCESSING of the PhotoPlethismoGraphic (PPG) signal (Normally the PPG signal in Pulse Oximeters is used only to compute heart rate and SpO2). The raw data is transferred from the watch oximeter to the smartphone using a standard Bluetooth protocol.

The Post-processing uses wavelet signal processing to estimate and display certain Hemodynamic parameters like Blood Pressure (BP) and Cardiac Output (CO) in a continuous and graphical way on a standard Android device. In addition to the standard heart rate and SpO2, the application displays the measured PPG signal and estimated continues BP and CO.

HeartBeat is the only device that can non-invasively estimate Continuous BP and its Cardiac Output component and the resistance component in a mobile wearable device. Differentiating between these 2 components can play a major role in helping the doctor to understand the effect of cardiovascular medications and Lifestyle interventions.

The trial will compare blood pressure and cardiac output parameters measured during Stress Echocardiography using an echo cardiograph and standard sphygmomanometer to the parameters generated by the application.

Trial goals

* Feasibility tests for the HeartBeat application as a tool for monitoring BP and CO changes over time
* Compare BP and CO parameters generated by the applications to the ones measured by standard non-invasive equipment during a Stress Echocardiography
* Calculate additional parameters such as stroke volume, systematic vascular resistance and cardiac index

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to an Stress Echocardiography test for cardiac diagnostics
* Male and Female
* Between 18 to 90 years old

Exclusion Criteria:

* Under the age of 18 or over 90 years old
* Patients in Shock
* Patients with Moderate or Severe valvular disease
* Patients with severe sepsis
* Inadequate jurisprudence patients
* Patients supported by Amines

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that are referred to the Stress Echocardiography test and are not in the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output | Change from Baseline in Cardiac Output at 30 minutes
  Measurement of Cardiac Output at the beginning and the end of the test (30 minutes)

SECONDARY OUTCOMES:
Blood Pressure | Change from Baseline in Systolic and Diastolic blood pressure at 30 minutes
Heart rate | Change from Baseline in heart rate at 30 minutes
  Measurement of Systolic and Diastolic blood pressure at the beginning and the end of the test

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Neuman, MD, Principal Investigator — Meir Health Facility
Locations (1):
- Meir Health Center, Kfar Saba, Israel